CLINICAL TRIAL: NCT03190434
Title: Pivotal Study of the AL-SENSE in Diagnosis Amniotic Fluid Leakage
Status: Completed | Type: Observational
Sponsor: Common Sense (Other)
Responsible Party: Sponsor
Other Study IDs: F-04-13-5.4; F-04-13-5.4 REV-5 (Other: COMMON SENSE); 20162402 (Registry Identifier: WIRB PRO NUM)
Record Dates: First submitted 2017-06-05; First posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2006-08

CONDITIONS: AMNIOTIC FLUID LEAKAGE

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — vaginal fluids
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- amniotic fluid: amniotic fluid identification by AL-SENSE product
  Interventions: Device: AL-SENSE

INTERVENTIONS:
Device: AL-SENSE — The AL-SENSE reacts differently when in contact with amniotic fluid than it does with urine. The indicator changes color to blue-green and fades back to yellow in case of urine and changes to stable blue-green in case of amniotic fluid.

SUMMARY:
This study is designed to demonstrate that the performance of the AL-SENSE developed by Common Sense Ltd. is safe and effective and can be used to indicate if the patient may be experiencing an amniotic fluid leakage or a "water breaking". The AL-SENSE is an extended shelf-life product that is technically simple, fast to react, visually readable, and therefore enables women to test the cause of any unidentified wetness. An additional, secondary objective is to show that the AL-SENSE is associated with levels of sensitivity and specificity that are comparable to those specified for the currently marketed AMNIOTESTTM (nitrazine yellow swabs; PRO LAB Diagnostics) product.

DETAILED DESCRIPTION:
Baseline/ Screening

Potential subjects may undergo the informed consent process in the outpatient clinic.

Subjects attending the labor and delivery unit of the hospital or emergency clinic and reporting unidentified wetness (undetermined whether this is amniotic fluid leakage or urinary incontinence) will be enrolled in this study. After informed consent is obtained, each subject will be given a single AL-SENSE to use up to 12 hours or until the perception of wetness. The clinician will explain the proper use and handling of the AL-SENSE and how to read the result. The participants will be provided with instructions for use and also directed to read the Instructions For Use (IFU) prior to applying the AL-SENSE pad.

Product Usage After usage, the subject will read and record any occurrence of color change of the AL-SENSE 10 minutes after the liner removal and to mark if it changes color to blue or to green or not on the designated form.. The used liner will be placed in a separate sealed envelope with the subject's ID and product name and protocol number on the outside.

The subjects will fill out the questionnaire regarding the product usage experience and the liner color reading with no help from the investigator, to validate IFU reading comprehension. The completed form will be placed in a sealed envelope with the subject's initials and study number on the outside.

Clinical Diagnosis A blinded clinician will perform a "standard clinical diagnosis" (clinical assessment), and record the results on a worksheet to be included in the case report form. The standard clinical diagnostic methods will include the following tests: (1) Pooling test, (2) Ferning test, (3) Nitrazine paper or pH paper test. A positive Pooling test and/or positive results in both the Nitrazine or pH test and the Ferning test will be defined as a positive clinical test result for amniotic fluid.

Although the preferred sequence is using the liner before clinical diagnosis, diagnostic procedures may be done before liner use, as long as lubricants are not used for procedures. The use of lubricants interferes with the accuracy of liner reaction to amniotic fluid.

If the liner is removed for clinical testing before sufficient fluid has collected, it may either be reused or a fresh liner may be dispensed. Note that any use of lubricants contraindicates further usage of Al-Sense.

The subject is expected to remain at the hospital for the duration of the test for completing the "standard clinical diagnosis" tests, required by the protocol.

A positive Pooling test or positive results in the other 2 tests is defined as a positive clinical assessment.

Although the performance of the AL-SENSE is examined in this study, subject treatment will be based only on the standard hospital diagnostic methods.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and 45 years.
* Subject minimum 16 weeks of pregnancy.
* Who will sign the informed consent form.
* Who arrive at the obstetric department reporting a feeling of vaginal wetness feeling undetermined whether this is amniotic fluid leakage or urinary incontinence).

Exclusion Criteria:

* Subject who has experienced intermittent vaginal bleeding between the 2nd and 3rd trimester.
* Subjects that have had sexual relations within the last 12 hours.
* Subject is unable or unwilling to cooperate with study procedures.
* Subject used the AL-SENSE before joining this study.
* Subject that has been diagnosed with Bacterial Vaginosis or Trichomonas infection within the last 3 days.
* Subject using vaginal products such as some douching formulas, some antibiotic treatments which reduce lactobacillus population.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women arriving at the hospital and reporting unidentified wetness
Sampling Method: Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2006-05; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
amniotic fluid leakage | day 1
  The primary efficacy endpoints are: presence or absence of a blue- green stain on a yellow background as observed by the subject yielded by the AL-SENSE in addition to the binary clinical diagnosis (positive/negative), in order to assess the sensitivity and specificity of the AL-SENSE versus the standard clinical diagnosis.

SECONDARY OUTCOMES:
result reading clarity | day 1
  The secondary endpoints of this study are: presence or absence of a blue-green stain on a yellow background as yielded by the AL-SENSE and observed by the clinician and a measurement of patient comfort while using AL-SENSE and reading the results. This will help demonstrate the ability of the subject to accurately interpret the AL-SENSE test results.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Black, MD, Principal Investigator — Ottawa Hospital Research Institute

IPD SHARING:
Plan to Share IPD: No